CLINICAL TRIAL: NCT05125679
Title: A Phase 4, Interventional, Single-arm, Open-label Study Evaluating the Effect of Guselkumab on Cardiovascular Risk Surrogate Markers in Participants With Moderate to Severe Plaque Psoriasis
Brief Title: Effect of Guselkumab on Cardiovascular Risk Surrogate Markers in Participants With Moderate to Severe Plaque Psoriasis
Acronym: G-CARE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated (A strategic decision was made not to further execute the study. This decision was not based on a safety concern)
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109033; 2020-004061-39 (EudraCT Number); CNTO1959PSO4015 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guselkumab (Experimental): Participants will receive guselkumab 100 milligrams (mg) by subcutaneous injection at Weeks 0, 4, 12, 20 and 28.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered by subcutaneous injection.

SUMMARY:
The purpose of this study is to evaluate the effect of guselkumab on coronary flow reserve (CFR), measured by transthoracic doppler-echocardiography, in participants with moderate-to-severe psoriasis and intermediate cardiovascular risk.

DETAILED DESCRIPTION:
Psoriasis is a common chronic inflammatory disease that affects 2 percent (%)-3% of the population and has an impact on physical and emotional health-related quality-of-life that is comparable to major illnesses such as cancer, heart disease and depression. Guselkumab is a fully human immunoglobulin G1 lambda monoclonal antibody that binds to the p19 protein subunit of human interleukin 23 (IL-23) with high specificity and affinity. Binding of guselkumab to the IL-23 p19 subunit blocks the binding of extracellular IL-23 to the cell surface IL-23 receptor, inhibiting IL-23 specific intracellular signaling and subsequent cytokine production. Guselkumab is indicated for the treatment of moderate-to-severe plaque psoriasis in adults who are candidates for systemic therapy. This study aims to investigate the efficacy of guselkumab in reducing surrogate parameters of vascular dysfunction and cardiovascular risk. This study will consist of two Screening Visits (Screening Visit S1 at a maximum of 2 weeks prior to Screening Visit S2, to occur at a minimum of 2 weeks and maximum of 4 weeks prior to Week 0), a Treatment Phase (up to 28 weeks), Final Efficacy Visit 4 weeks later (Week 32), and Final Safety Visit (Week 40). The efficacy assessments will be done locally at the sites and safety will be monitored by assessment of adverse events, clinical laboratory tests, physical examinations, vital signs, and concomitant medication review. The total duration of the study will be 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of moderate-to-severe plaque psoriasis (with or without psoriatic arthritis [PsA]) for at least 6 months prior to the first dose of guselkumab at Week 0. Moderate-to-severe plaque psoriasis is defined as having a psoriasis area and severity index (PASI) score greater than or equal to (>=) 12, investigator global assessment (IGA) score >= 3 and involved body surface area (BSA) >= 10 percent (%) at Screening Visit S1
* The participant has intermediate cardiovascular risk defined as having a coronary flow reserve (CFR) score >= 2 to less than or equal to (<=) 3.5 (criterion to be assessed by cardiologist at Screening Visit S2 and Week 0)
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at Screening Visit S1
* Within 2 months before the first administration of guselkumab, the participant has a negative QuantiFERON-TB Gold test result, or has a newly identified positive QuantiFERON-TB Gold test result in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated before the first administration of guselkumab
* The participant has a chest radiograph (posterior-anterior view), taken within 3 months before the first administration of study agent and read by a qualified radiologist, with no evidence of current, active tuberculosis (TB) or old, inactive TB

Exclusion Criteria:

* The participant has a predominantly non-plaque form of psoriasis (example, erythrodermic, guttate, or pustular)
* The participant has uncontrolled hypertension that needs immediate medical attention (criterion to be assessed by the dermatologist at Screening Visit S1 and by the cardiologist at Screening Phase 2)
* The participant has taken any prohibited therapies before the planned first dose of guselkumab
* A female participant is pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or within 5 months after the last dose of guselkumab
* The participant has any clinically significant evidence of cardiac functional or valvular abnormalities, other than intermediate cardiovascular risk defined by CFR score >=2 and <=3.5, observed during the CFR assessment (criterion to be assessed by the dermatologist at Screening Visit S1, and to be confirmed by the cardiologist at Screening Visit S2)
* The participant has any contraindications to adenosine infusion, or other contraindications listed in the summary of product characteristics (SmPC) (criterion to be assessed by the dermatologist at Screening Visit S1 and confirmed by the cardiologist at Screening Visit S2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (5):
- Germany (2):
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitatsklinikum Leipzig AOR, Leipzig
- Attikon Hospital, Athens, Greece
- Italy (2):
  - Ospedale San Giovanni di Dio, Cagliari
  - Azienda Ospedaliera di Padova, Padua

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 adult participants diagnosed with moderate-to-severe plaque psoriasis (with or without psoriatic arthritis) for at least 6 months prior to the first dose of guselkumab at Week 0 (baseline) of the study entry were enrolled and treated with at least one dose of guselkumab.
Groups:
- Guselkumab 100 mg: Nicotine Users: Participants who were nicotine users (who had used tobacco products and/or nicotine products) received guselkumab 100 milligrams (mg) subcutaneous (SC) injection at Weeks 0, 4, 12, 20, and 28.
- Guselkumab 100 mg: Non-Nicotine Users: Participants who were non-nicotine users (who had refrained from using tobacco/nicotine products for at least 3 months prior to screening visit 1 [4 to 6 weeks prior to Week 0]) received guselkumab 100 mg SC injection at Weeks 0, 4, 12, 20, and 28.
Period: Overall Study
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Started | 7 | 8
Participants With Intermediate Cardiovascular Risk (ICR) (Participants who had CFR value greater than or equal to (>=) 2 and less than or equal to (<=) 3.5 at screening Visit 2 and at Week 0.) | 3 | 5
Completed | 5 | 3
Not Completed | 2 | 5
Not completed — Study Terminated by Sponsor | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (14.09) | 39.1 (12.8) | 44.1 (14.06)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 6 | 8 | 14
  From 65 to 84 years | 1 | 0 | 1
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Coronary Flow Reserve (CFR) at Week 32
Description: Change from baseline in CFR at Week 32 were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 micrograms per kilogram per minute (mcg/kg/min; coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest.
Time Frame: Baseline (Week 0) and Week 32
Population: FAS included all participants who received at least 1 dose of guselkumab. Here, 'N' (number of participants analyzed) signifies number of treated participants evaluable for this outcome measure with ICR defined by CFR >=2 and <=3.5 at screening visit 2 (2 to 4 weeks prior to Week 0) and baseline (Week 0).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 3
ratio | -0.080 (0.2773) | 0.173 (0.6478)

2. Secondary Outcome: Change From Baseline in CFR at Week 16
Description: Change from baseline in CFR at Week 16 were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 mcg/kg/min (coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest.
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 2
ratio | 0.113 (0.3099) | 0.435 (0.2899)

3. Secondary Outcome: Change From Baseline in Absolute Global Longitudinal Strain (GLS) at Week 16
Description: Change from baseline in absolute GLS at Week 16 were reported. GLS is a myocardial deformation analysis that predominantly reflects the function of sub-endocardial longitudinally oriented fibers, which are most prone to ischemic damage and wall stress. The GLS is calculated at systole and diastole. Speckle tracking echocardiography (STE) were employed for the detection of left-ventricular (LV) myocardial strain. GLS is a measure of longitudinal shortening of the myocardium as a percentage (change in length as a proportion to baseline length), thus explaining the negative values.
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of myocardial shortening
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 2
percentage of myocardial shortening | -1.377 (0.9660) | -2.625 (0.9829)

4. Secondary Outcome: Change From Baseline in Absolute GLS at Week 32
Description: Change from baseline in absolute GLS is a myocardial deformation analysis that predominantly reflects the function of sub-endocardial longitudinally oriented fibers, which are most prone to ischemic damage and wall stress. The GLS is calculated at systole and diastole. Speckle tracking echocardiography (STE) were employed for the detection of left-ventricular (LV) myocardial strain. GLS is a measure of longitudinal shortening of the myocardium as a percentage (change in length as a proportion to baseline length), thus explaining the negative values.
Time Frame: Baseline (Week 0) and Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of myocardial shortening
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 3
percentage of myocardial shortening | 0.850 (0.6065) | -3.063 (3.0593)

5. Secondary Outcome: Change From Baseline in Carotid-femoral Pulse Wave Velocity (cfPWV) at Week 16
Description: Change from baseline in cfPWV at Week 16 were reported. cfPWV is a direct measurement, and the most simple, non-invasive, robust, and reproducible method to determine arterial stiffness. cfPWV was determined from the time taken for the arterial pulse to propagate from the carotid to the femoral artery. cfPWV was calculated as cfPWV = distance (meters) / transit time (seconds).
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter per second (m/s)
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 2
meter per second (m/s) | 0.77 (0.503) | -0.35 (0.495)

6. Secondary Outcome: Change From Baseline in cfPWV at Week 32
Description: Change from baseline in cfPWV at Week 32 were reported. cfPWV is a direct measurement, and the most simple, non-invasive, robust, and reproducible method to determine arterial stiffness. cfPWV was determined from the time taken for the arterial pulse to propagate from the carotid to the femoral artery. cfPWV was calculated as cfPWV = distance (meters) / transit time (seconds).
Time Frame: Baseline (Week 0) and Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter per second (m/s)
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 2
meter per second (m/s) | 1.37 (1.332) | -1.00 (0.283)

7. Secondary Outcome: Change From Baseline in CFR at Week 16 Among Participants With CFR >=2 to Less Than (<) 2.75 at Baseline
Description: Change from baseline in CFR at Week 16 among participants with CFR >=2 to <2.75 at baseline were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 mcg/kg/min (coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest
Time Frame: Baseline (Week 0) and Week 16
Population: FAS included all participants who received at least 1 dose of guselkumab. Here, 'N' (number of participants analyzed) signifies number of treated participants evaluable for this outcome measure with ICR defined by CFR >=2 to <2.75 at baseline (Week 0). None of the nicotine users had the baseline CFR measurement of >=2 to <2.75 and thus, no data was reported for arm 'Guselkumab 100 mg: Nicotine Users'.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 0 | 2
ratio |  | 0.435 (0.2899)

8. Secondary Outcome: Change From Baseline in CFR at Week 32 Among Participants With CFR >=2 to <2.75 at Baseline
Description: Change from baseline in CFR at Week 32 among participants with CFR >=2 to <2.75 at baseline were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 mcg/kg/min (coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest
Time Frame: Baseline (Week 0) and Week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 0 | 3
ratio |  | 0.173 (0.6478)

9. Secondary Outcome: Change From Baseline in CFR at Week 16 Among Participants With CFR >=2.75 to <=3.5 at Baseline
Description: Change from baseline in CFR at Week 16 among participants with CFR >=2.75 to <=3.5 at baseline were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 mcg/kg/min (coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest
Time Frame: Baseline (Week 0) and Week 16
Population: FAS included all participants who received at least 1 dose of guselkumab. Here, 'N' (number of participants analyzed) signifies number of treated participants evaluable for this outcome measure with ICR defined by CFR >=2.75 to <=3.5 at baseline (Week 0). None of the non-nicotine users had the baseline CFR measurement of >=2.75 to <=3.5 and thus, no data was reported for arm 'Guselkumab 100 mg: Non-Nicotine Users'.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 0
ratio | 0.113 (0.3099) |

10. Secondary Outcome: Change From Baseline in CFR at Week 32 Among Participants With CFR >=2.75 to <=3.5 at Baseline
Description: Change from baseline in CFR at Week 32 among participants with CFR >=2.75 to <=3.5 at baseline were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 mcg/kg/min (coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest
Time Frame: Baseline (Week 0) and Week 32
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 3 | 0
ratio | -0.080 (0.2773) |

11. Secondary Outcome: Change From Baseline in CFR Among Nicotine Users and Non-nicotine Users at Weeks 16
Description: Change from baseline in CFR among nicotine users and non-users at Week 16 were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 mcg/kg/min (coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest
Time Frame: Baseline (Week 0) and Week 16
Population: FAS included all participants who received at least 1 dose of guselkumab. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Guselkumab 100 mg (Nicotine Users): Participants who were nicotine users (who had used tobacco products and/or nicotine products) received guselkumab 100 mg SC injection at Week 0, 4, 12, 20 and 28.
- Guselkumab 100 mg (Non-Nicotine Users): Participants who were non-nicotine users (who had refrained from using tobacco/nicotine products for at least 3 months prior to baseline [Week 0]) received guselkumab 100 mg SC injection at Week 0, 4, 12, 20, and 28.
Arm/Group | Guselkumab 100 mg (Nicotine Users) | Guselkumab 100 mg (Non-Nicotine Users)
Number analyzed (Participants) | 5 | 5
ratio | 0.024 (0.6124) | 0.132 (0.7874)

12. Secondary Outcome: Change From Baseline in CFR Among Nicotine Users and Non-nicotine Users at Weeks 32
Description: Change from baseline in CFR among nicotine users and non-nicotine users at Weeks 32 were reported. CFR was described as ability of coronary blood flow to increase substantially when required by metabolic demands, which might be up to 4 to 5 times greater during normal exercise compared to resting, and even greater with administration of pharmacological agents. CFR was measured non-invasively using transthoracic doppler echocardiography. First, initial spectral Doppler signals in distal portion of left anterior descending artery (LAD) was recorded and then adenosine 140 mcg/kg/min (coronary vasodilator) was administered for 5 minutes. Doppler signals were recorded continuously during the period of adenosine infusion. Baseline (Week 0): last non-missing measurement prior to or on day of 1st dose of guselkumab. CFR is the ratio of blood flow at stress during maximal dilation of the coronary arteries to blood flow at rest
Time Frame: Baseline (Week 0) and Week 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Guselkumab 100 mg (Nicotine Users) | Guselkumab 100 mg (Non-Nicotine Users)
Number analyzed (Participants) | 6 | 6
ratio | 0.487 (1.1418) | -0.253 (0.7173)

13. Secondary Outcome: Change From Baseline in Absolute GLS Among Nicotine Users and Non-users at Week 16
Description: Change from baseline in absolute GLS among nicotine users and non-nicotine users at Week 16 were reported. GLS is a myocardial deformation analysis that predominantly reflects the function of sub-endocardial longitudinally oriented fibers, which are most prone to ischemic damage and wall stress. The GLS is calculated at systole and diastole. Speckle tracking echocardiography (STE) were employed for the detection of left-ventricular (LV) myocardial strain. GLS is a measure of longitudinal shortening of the myocardium as a percentage (change in length as a proportion to baseline length), thus explaining the negative values.
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of myocardial shortening
Arm/Group | Guselkumab 100 mg (Nicotine Users) | Guselkumab 100 mg (Non-Nicotine Users)
Number analyzed (Participants) | 5 | 4
percentage of myocardial shortening | -1.496 (0.8452) | -0.780 (2.3553)

14. Secondary Outcome: Change From Baseline in Absolute GLS Among Nicotine Users and Non-users at Week 32
Description: Change from baseline in absolute GLS among nicotine users and non-nicotine users at Week 32 were reported. GLS is a myocardial deformation analysis that predominantly reflects the function of sub-endocardial longitudinally oriented fibers, which are most prone to ischemic damage and wall stress. The GLS is calculated at systole and diastole. Speckle tracking echocardiography (STE) were employed for the detection of left-ventricular (LV) myocardial strain. GLS is a measure of longitudinal shortening of the myocardium as a percentage (change in length as a proportion to baseline length), thus explaining the negative values.
Time Frame: Baseline (Week 0) and Week 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of myocardial shortening
Arm/Group | Guselkumab 100 mg (Nicotine Users) | Guselkumab 100 mg (Non-Nicotine Users)
Number analyzed (Participants) | 6 | 5
percentage of myocardial shortening | -0.060 (2.2065) | -2.490 (2.3020)

15. Secondary Outcome: Change From Baseline in cfPWV Among Nicotine Users and Non-users at Week 16
Description: Change from baseline in cfPWV among nicotine users and non-nicotine users at Week 16 were reported. cfPWV is a direct measurement, and the most simple, non-invasive, robust, and reproducible method to determine arterial stiffness. cfPWV was determined from the time taken for the arterial pulse to propagate from the carotid to the femoral artery. cfPWV was calculated as cfPWV= distance (meters)/ transit time (seconds).
Time Frame: Baseline (Week 0) and Week 16
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: meter per second (m/s)
Arm/Group | Guselkumab 100 mg (Nicotine Users) | Guselkumab 100 mg (Non-Nicotine Users)
Number analyzed (Participants) | 5 | 4
meter per second (m/s) | 0.34 (0.716) | -0.38 (0.330)

16. Secondary Outcome: Change From Baseline in cfPWV Among Nicotine Users and Non-users at Week 32
Description: Change from baseline in cfPWV among nicotine users and non-nicotine users at Week 32 were reported. cfPWV is a direct measurement, and the most simple, non-invasive, robust, and reproducible method to determine arterial stiffness. cfPWV was determined from the time taken for the arterial pulse to propagate from the carotid to the femoral artery. cfPWV was calculated as cfPWV= distance (meters)/ transit time (seconds).
Time Frame: Baseline (Week 0) and Week 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: meter per second (m/s)
Arm/Group | Guselkumab 100 mg (Nicotine Users) | Guselkumab 100 mg (Non-Nicotine Users)
Number analyzed (Participants) | 5 | 5
meter per second (m/s) | 0.84 (1.191) | -0.80 (0.791)

17. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An adverse event (AE) was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Any AE occurring at or after initial administration study intervention (guselkumab) through the day of last dose within the study phase plus 12 weeks or the date of the Final Safety visit, whichever was the latest, was considered to be TEAE.
Time Frame: Week 0 up to 12 weeks post last dose of study drug (up to Week 40)
Population: The safety analysis set included all participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
Number analyzed (Participants) | 7 | 8
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Week 0 up to 12 weeks post last dose of study drug (up to Week 40)
Description: The safety analysis set included all participants who received at least 1 dose of guselkumab.
Arm/Group | Guselkumab 100 mg: Nicotine Users | Guselkumab 100 mg: Non-Nicotine Users
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/8
Other Adverse Events (participants affected / at risk) | 1/7 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guselkumab 100 mg: Nicotine Users (N=7) | Guselkumab 100 mg: Non-Nicotine Users (N=8)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guselkumab 100 mg: Nicotine Users (N=7) | Guselkumab 100 mg: Non-Nicotine Users (N=8)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Sponsor terminated the study solely due to lack of enrolment. Due to small number of enrolled participants, it was not possible to evaluate the primary or secondary objectives for this study as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. If requested by the Sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT05125679/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT05125679/SAP_001.pdf